CLINICAL TRIAL: NCT00004533
Title: Phase I Randomized Study of Adeno-Associated Virus-CFTR Vector in Patients With Cystic Fibrosis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Collaborators: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: 199/14137; UF-G-037-1996 (Other: University of Florida); TGC-AAV-9502; P01DK058327 (NIH); R01DK051809 (NIH)
Record Dates: First submitted 2000-01-28; First posted 2000-01-31 (Estimated); Last update posted 2017-06-01 (Actual); Status verified 2017-05

CONDITIONS: Cystic Fibrosis
Keywords: cardiovascular and respiratory diseases; cystic fibrosis; genetic diseases and dysmorphic syndromes; rare disease
MeSH Terms: conditions — Cystic Fibrosis; Respiratory Tract Diseases; Genetic Diseases, Inborn; Rare Diseases

INTERVENTIONS:
Drug: Adeno-associated virus-CFTR vector

SUMMARY:
OBJECTIVES:

I. Determine the maximum tolerated dose of recombinant adeno-associated virus-CFTR vector in patients with cystic fibrosis.

II. Assess the safety of this gene therapy in these patients.

III. Assess the in vivo gene transfer of this vector in these patients.

IV. Assess the CFTR gene expression and physiologic activity following gene transfer in these patients.

V. Assess the clinical impact of CFTR gene expression following gene transfer in these patients.

VI. Monitor patient immune response directed against CFTR or vector components following vector administration.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE:

This is a randomized, dose escalation, double blind, placebo controlled, multicenter study. Patients are randomized to receive either adeno-associated virus-CFTR (AAV-CFTR) vector or placebo.

Patients undergo tests on days -10 to -4 to rule out adenovirus and adeno-associated virus infections. Patients then receive AAV-CFTR vector intranasally to the right or left inferior turbinates and placebo to the other side of the nose. The next day, patients receive an endobronchial dose of AAV-CFTR vector to the superior segment of the right lower lobe.

Cohorts of 2-4 patients each receive escalating doses of AAV-CFTR vector until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose level immediately preceding the dose at which at least 2 subjects develop dose limiting toxicity.

Patients are followed at day 10, then at 1, 2, 3, 6, 9, and 12 months.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics--

Diagnosis of cystic fibrosis (CF) with mild to moderate lung disease; FVC at least 60% predicted; Schwachman-Kulczycki score at least 65; Sweat chloride greater than 60 mEq/L

All CF genotypes allowed

No sputum colonization with Burkholderia cepacia or another multiply resistant organism

No recurrent or intermittent hemoptysis; At least 1 year since significant hemoptysis requiring transfusion or embolization OR Coughing of greater than 30 mL of blood more often than once a week

--Prior/Concurrent Therapy--

At least 30 days since hospitalization or home intravenous antibiotic therapy for pulmonary exacerbation

No concurrent investigational drugs or therapy

--Patient Characteristics--

Other: No concurrent cigarette smoking; Not pregnant or nursing; Negative pregnancy test; Fertile patients must use effective contraception

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 19
Dates: Start 1999-08; Primary Completion 2002-08 (Actual); Study Completion 2002-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Terence Flotte, Study Chair — University of Florida

REFERENCES:
- [Result] Flotte TR, Zeitlin PL, Reynolds TC, Heald AE, Pedersen P, Beck S, Conrad CK, Brass-Ernst L, Humphries M, Sullivan K, Wetzel R, Taylor G, Carter BJ, Guggino WB. Phase I trial of intranasal and endobronchial administration of a recombinant adeno-associated virus serotype 2 (rAAV2)-CFTR vector in adult cystic fibrosis patients: a two-part clinical study. Hum Gene Ther. 2003 Jul 20;14(11):1079-88. doi: 10.1089/104303403322124792. PMID 12885347